CLINICAL TRIAL: NCT03351504
Title: Solar Lighting Intervention Trial to Reduce Indoor Air Pollution and Improve Adult Respiratory Health in Rural Uganda
Brief Title: Solar Lighting to Reduce Indoor Air Pollution in Rural Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Peggy S Lai, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000306/PHS
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2020-12

CONDITIONS: Pollution; Exposure; Hypertension; Pollution Related Respiratory Disorder
Keywords: household air pollution; fine particulate matter; kerosene
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed using dummy codes to represent intervention and control groups by an independent statistician; blinding of the intervention to the participants and field team is not possible, but data analysis will take place prior to unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (usual lighting) (No Intervention): Participants will continue to use their usual lighting sources.
- Intervention (solar lighting) (Experimental): Participants will receive an indoor solar lighting system
  Interventions: Other: Solar lighting system

INTERVENTIONS:
Other: Solar lighting system — consisting of a solar panel, rechargeable lead acid battery, charge controller, wiring and switches to 4 lighting points fitted with LED bulbs. This system will include a two-year service warranty.
  Arms: Intervention (solar lighting)

SUMMARY:
This study evaluates the impact of a solar lighting system on kerosene lamp use, levels of indoor air pollution, and health in women living in rural Uganda. Half of the participants will receive the lighting systems immediately, while the other half will receive them after an 18 month delay.

DETAILED DESCRIPTION:
One fifth of the global population relies on kerosene lamps for lighting, yet few studies have focused on kerosene lighting as a source of indoor air pollution. In our preliminary studies performed in Uganda, we show that homes using solar lighting have much lower levels of indoor air pollution compared to homes using kerosene lighting. The primary goal of this study is to determine the extent to which solar lighting will reduce kerosene use and indoor air pollution in rural Uganda, whether this intervention improves lung health, and to identify the role bacteria in our gut have on determining whether or not people will get sick from indoor air pollution.

ELIGIBILITY:
Inclusion Criteria:

* Women living in Nyakabare Parish, Uganda with no prior history of chronic lung disease

Exclusion Criteria:

* Current active tuberculosis in any family member

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Fine particulate matter (PM2.5) and Black Carbon | 48 hour
  Sampling for PM2.5 and Black Carbon over 48 hours will be collected

SECONDARY OUTCOMES:
Daily use of solar lighting system (hours per day) | baseline, 3 months, 6 months, 12 months after the intervention
  A current monitory is installed as part of the solar lighting system that measures the hours per day each light switch is turned on
Blood pressure | baseline, 3 months, 6 months, 12 months after the intervention
  Resting blood pressure
Forced Expiratory Volume in one Second (FEV1) | baseline, 3 months, 6 months, 12 months after the intervention
  Pre- and Post- bronchodilator spirometry
Heart rate variability | baseline, 3 months, 6 months, 12 months after the intervention
  Resting 10 minute heart rate variability
Stool microbiome | baseline, 3 months, 6 months, 12 months after the intervention
  Microbial sequencing of the stool will be performed
Qualitative interviews | Post-intervention
  1:1 qualitative interviews will be performed with participants
Respiratory symptoms | baseline, 3 months, 6 months, 12 months after intervention
  Presence/absence of respiratory symptoms based on the American Thoracic Society Respiratory Disease questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peggy S Lai, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CY, Nuwagira E, Tisza M, Kim M, Tayebwa M, Vieira J, Lam N, Wallach E, Wiens M, Tsai AC, Valeri L, Vallarino J, Allen JG, Lai PS. Effect of household air pollution on the gut microbiome and virome of adult women living in Uganda. Environ Health Perspect. 2025 May 21. doi: 10.1289/EHP16002. Online ahead of print. PMID 40397799
- [Derived] Ponticiello M, Nuwagira E, Tayebwa M, Mugerwa J, Nahabwe H, Nakasita C, Tumuhimbise JB, Lam NL, Wiens MO, Vallarino J, Allen JG, Muyanja D, Tsai AC, Sundararajan R, Lai PS. "If you have light, your heart will be at peace": A qualitative study of household lighting and social integration in southwestern Uganda. J Glob Health. 2023 Apr 14;13:04026. doi: 10.7189/jogh.13.04026. PMID 37052216
- [Derived] Wallach ES, Lam NL, Nuwagira E, Muyanja D, Tayebwa M, Valeri L, Tsai AC, Vallarino J, Allen JG, Lai PS. Effect of a solar lighting intervention on fuel-based lighting use and exposure to household air pollution in rural Uganda: A randomized controlled trial. Indoor Air. 2022 Feb;32(2):e12986. doi: 10.1111/ina.12986. PMID 35225388